CLINICAL TRIAL: NCT06630494
Title: A Single-center, Single-arm, Open-label, Single-dose Phase I Clinical Study to Evaluate Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of rhTPO in Healthy Caucasian Participants. Approximately 22 Subjects Will be Enrolled.
Brief Title: Phase I Study to Evaluate rhTPO in Healthy Caucasian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 3SBIO AU PTY LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: rhTPO-101-AUS
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subjects
Keywords: rhTPO
MeSH Terms: interventions — Thrombopoietin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Caucasian volunteers (Experimental): Single abdominal subcutaneous injection of the study drug will be given on D1. The administration and follow-up observation period will be 29 days (D1~D29). Participants may be discharged at D7 at the judgment of the investigator. PK blood samples will be collected from D-1 to D14, tolerance and safety will be observed from D1 to D29, and blood samples for PD and anti-drug antibody (ADA) will be collected from screening to D29. After completion of relevant assessments on D29, participants will be considered as having completed this study.
  Interventions: Drug: Recombinant human thrombopoietin for injection (rhTPO)

INTERVENTIONS:
Drug: Recombinant human thrombopoietin for injection (rhTPO) — Single abdominal subcutaneous injection of the study drug will be given on D1. The administration and follow-up observation period will be 29 days (D1~D29). Participants may be discharged at D7 at the judgment of the investigator. PK blood samples will be collected from D-1 to D14, tolerance and safety will be observed from D1 to D29, and blood samples for PD and anti-drug antibody (ADA) will be collected from screening to D29. After completion of relevant assessments on D29, participants will be considered as having completed this study.

SUMMARY:
This is a single-center, single-arm, open-label, single-dose phase I clinical study to evaluate pharmacokinetics (PK), pharmacodynamics (PD), safety and tolerability of Recombinant Human Thrombopoietin for Injection (rhTPO) in healthy Caucasian participants. Approximately 22 healthy Caucasian participants will be enrolled for this study.

One dose level is planned in this study, and participants will receive a single abdominal subcutaneous injection at a dose of 300 U/kg after entering the study.

Participants will undergo screening, admission (baseline), administration and follow-up observation period. Participants will sign an informed consent form before any study procedures are performed. During screening, all participants will be screened for study eligibility within 28 days prior to administration. Eligible participants will be admitted to the clinical study ward no later than one day prior to dosing (D-1). Participants need to fast for at least 10 hours prior to dosing and 4 hours after dosing. Single abdominal subcutaneous injection of the study drug will be given on D1. The administration and follow-up observation period will be 29 days (D1~D29). Participants may be discharged at D7 at the judgment of the investigator. PK blood samples will be collected from D-1 to D14, tolerance and safety will be observed from D1 to D29, and blood samples for PD and ADA will be collected from screening to D29. After completion of relevant assessments on D29, participants will be considered as having completed this study.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label, single-dose phase I clinical study to evaluate pharmacokinetics, pharmacodynamics, safety and tolerability of Recombinant Human Thrombopoietin for Injection (rhTPO) in healthy Caucasian participants. Approximately 22 healthy Caucasian participants will be enrolled for this study.

One dose level is planned in this study, and participants will receive a single abdominal subcutaneous injection at a dose of 300 U/kg after entering the study.

Participants will undergo screening, admission (baseline), administration and follow-up observation period. Participants will sign an informed consent form before any study procedures are performed. During screening, all participants will be screened for study eligibility within 28 days prior to administration. Eligible participants will be admitted to the clinical study ward no later than one day prior to dosing (D-1). Participants need to fast for at least 10 hours prior to dosing and 4 hours after dosing. Single abdominal subcutaneous injection of the study drug will be given on D1. The administration and follow-up observation period will be 29 days (D1~D29). Participants may be discharged at D7 at the judgment of the investigator. PK blood samples will be collected from D-1 to D14, tolerance and safety will be observed from D1 to D29, and blood samples for PD and ADA will be collected from screening to D29. After completion of relevant assessments on D29, participants will be considered as having completed this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

  1. Healthy Caucasian adult male and female participants aged 18-50 years (inclusive) at the time of informed consent. Caucasian is defined as of European, Middle Eastern, or North African descent.
  2. Male participants weighing no less than 50 kg. Female participants should not weigh less than 45 kg.
  3. Body mass index (BMI) within the range 18.0 to 32.0 kg/m2 (inclusive). Note: BMI = weight [kg] / (height [m])2
  4. Participants are in good general health as determined by the investigator, based on a medical evaluation including medical history, vital signs, physical examination, 12-lead electrocardiogram, clinical safety laboratory tests; Note: Any results outside of the reference range at screening or baseline may be repeated once per the Investigator's discretion for the purpose of further determining eligibility.
  5. Platelet counts must be within the normal range; measurements can repeat once for verification, if necessary.
  6. Women of childbearing potential (WOCBP, see section 5.3.3) must have a negative serum or urine pregnancy test prior to the start of study drug and must not be breastfeeding, lactating or planning pregnancy during the study period. WOCBP who are not exclusively in same-sex relationships and males with partners of child-bearing potential must agree to use adequate contraception from signing the informed consent until 3 months after completion of the study. In addition, females must not donate ova (eggs) and males must not donate sperm from signing the informed consent until 3 months after completion of the study;
  7. Negative for COVID-19 based on the nasopharyngeal or oropharyngeal swab with the method of real-time reverse transcription-polymerase chain reaction (RT-PCR) at Screening and Day-1.
  8. Volunteer to participate in this study, be able to understand and comply with the clinical study protocol requirements, and sign the informed consent form in writing.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  1. History of hypersensitivity to components of study drug or analogs; history of anaphylaxis or other significant allergy in opinion of the investigators.
  2. Known allergy to heparin or history of heparin-induced thrombocytopenia;
  3. Received a platelet transfusion within 2 weeks or platelet-boosting medication within 4 weeks prior to dosing;
  4. History of hospitalization or surgical procedure within 3 months prior to dosing, or bleeding from trauma or internal bleeding greater than 100 mL, or donating more than 100 mL of blood;
  5. History or presence of autoimmune disease, malignancy, thromboembolic disease, bleeding disorders, cardiovascular, hepatic, renal, muscular, hematopoietic, respiratory, neurological, or psychiatric disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, constituting a risk to the participant when taking the study drug; or interfering with the interpretation of data judged by the investigator; Note: Uncomplicated cholecystectomy and appendectomy are permitted; History of fully resolved childhood asthma is not permitted.
  6. History or presence of chronic diseases such as hypertension and diabetes (including type 1 and type 2 diabetes);
  7. History of malignancy with the exception of successfully treated basal cell or squamous cell skin cancer with no evidence of recurrence for 5 years.
  8. History of platelet clumping that prevents reliable measurement of platelet counts;
  9. Positive for Hepatitis B surface antigen (HBsAg), Hepatitis C Virus (HCV) antibody and Human Immunodeficiency Virus (HIV) antibody, Syphilis antibody; Note: Participants with positive hepatitis C antibody can be enrolled if a confirmatory negative hepatitis C RNA test is obtained.
  10. Immunization with a Corona Virus Disease 2019 (COVID-19) vaccine 14 days prior to dosing or planned vaccination within 30 days after dosing
  11. Use of prescription medication within 14 days prior to dosing and 7 days prior to dosing for over the counter medication/vitamins/herbal supplements (with the exception of contraception, occasional paracetamol < 2g/day, and standard dose of multivitamins).
  12. Consumption of alcohol, caffeinated products (coffee, tea, cola, chocolate), grapefruit fruits, or products containing grapefruit within 48 hours prior to dosing;
  13. Consumption of any poppy seeds (e.g., orange and poppy seed muffin, poppy seed bread) within 48 hours prior to screening and admission.
  14. History of drug abuse within 2 years prior to dosing; or positive alcohol/urine drug screen prior to dosing; Regular alcohol consumption within 6 months prior to dosing, i.e., on average more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits at 40% alcohol by volume or 150 mL of wine);
  15. Use of tobacco or nicotine products equivalent to more than 2 cigarettes a day on average within 3 months prior to dosing;
  16. Have special dietary requirements and are unable to comply with the diet offered and the corresponding regulations;
  17. Pregnant or breastfeeding female, or positive pregnancy test;
  18. Individuals who cannot tolerate venipuncture or who suffer from needle and blood sickness;
  19. Participation in another clinical study of investigational drug within 3 months prior to dosing;
  20. Other participants judged by the investigator to be unsuitable for participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Serum rhTPO concentration | pre-dosing and 14 days after dosing
  Pharmacokinetic index

CONTACTS AND LOCATIONS:
Overall Officials: Arockiaa Philo Aarthy Joseph, Ph.D, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network Pty Ltd., Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT06630494/Prot_000.pdf